CLINICAL TRIAL: NCT06589128
Title: Efficacy of Investigator Product for the Amelioration of Digital Eye Strain in Children: a Randomized, Double-blind, Placebo-controlled Human Clinical Trial
Brief Title: Efficacy of Investigator Product for the Amelioration of Digital Eye Strain in Children
Acronym: DES
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Dr. Lee Lai Kuan, Principal Investigator, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: USM-Astaxanthin-02/2024; R378 (Other Grant/Funding Number: Universiti Sains Malaysia)
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Digital Eye Strain (DES)
Keywords: Children; Digital Eye Strain; Astaxanthin
MeSH Terms: interventions — astaxanthine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Astaxanthin (Active Comparator): Oral astaxanthin supplement
  Interventions: Dietary Supplement: Astaxanthin Oral Capsule
- Placebo (Placebo Comparator): Oral placebo supplement
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Astaxanthin Oral Capsule — Once daily supplementation of oral astaxanthin capsule for 24 weeks
  Arms: Astaxanthin
Dietary Supplement: Placebo — Once daily supplementation of olive oil capsule for 24 weeks
  Arms: Placebo

SUMMARY:
Computer vision syndrome (CVS), also referred to as Digital eye strain (DES), is a group of eye and vision problems caused by prolonged use of electronic devices. The American Optometric Association (APA) defines DES as a group of eye and vision-related problems caused by prolonged computer, tablet, e-reader, and cell phone use. Currently, for more than 20 years, DES has been recognised as a public health issue, and the terms DES are also used to describe the condition, attributed to the wide range of digital devices associated with potential problems.

DETAILED DESCRIPTION:
Digital device usage has increased substantially in recent years across all age groups, so that extensive daily use for both social and professional purposes is now normal. Digital eye strain (DES), also known as computer vision syndrome, encompasses a range of ocular and visual symptoms, and estimates suggest its prevalence may be 50% or more among computer users. Symptoms fall into two main categories: those linked to accommodative or binocular vision stress, and external symptoms linked to dry eye. Although symptoms are typically transient, they may be frequent and persistent, and have an economic impact when vocational computer users are affected.

Astaxanthin is a naturally occurring red carotenoid pigment belonging to the family of xanthophylls, and is typically found in marine environments, especially in microalgae and seafood such as salmonids, shrimps and lobsters. Application fields of astaxanthin range from the food coloring industry, for its natural intense red color brightness, to aquaculture and poultry industries for its natural feed addictive properties. Due to its unique molecular structure, astaxanthin features some important biologic properties, mostly represented by strong antioxidant, anti-inflammatory and antiapoptotic activities. A growing body of evidence suggests that astaxanthin is efficacious in the prevention and treatment of several ocular diseases, ranging from the anterior to the posterior pole of the eye. In particular, astaxanthin seems to be effective in improving blood capillary circulation of the eyes. In Japan, human clinical trial showed that consuming 9mg of astaxanthin daily over four weeks significantly improved the eyes' ability to accommodate different focuses and reduce eye strain, hazy vision, flickering images, shoulder or back stiffness as compared to the control group. Astaxanthin has been reported to have an ocular accommodation improvement effect, and acts as a substance to help with asthenopia recovery and could contribute to the improvement of blood circulation in peripheral systems. Due to the well-known effects of helping 2 eyes in many ocular structures, astaxanthin is a superlative bodyguard to prevent smartphone eye damages.

DES is the most common eye problem associated with prolonged digital device use, characterized by symptoms such as dry eyes, itching, foreign body sensation, watering, blurring of vision, and headaches. It is increasingly common for present day children have grown up with electronic devices and this has become the norm in many of the more affluent societies. Some caregivers may even use such electronic technology as an "electronic pacifier" to calm and entertain their kids. Digital technology always raises concerns about a potential negative impact on the physical, cognitive, emotion and social well-being of the children. There is evidence that excessive screen time is associated with a variety of health harms among children, with evidence strongest for an unhealthy diet, adiposity, depressive symptoms and quality of life.

DES in children is of particular concerning, as it does not have any suggested medical treatment to ameliorate the symptoms. The role of nutrition as complementary medicine is getting scientific attention nowadays. Astaxanthin, a potent antioxidant classified under the red-pigment carotenoid, is a promising vision enhancer with numerous human clinical trial evidences conducted among the adults. However, limited research has been conducted to determine the effect of astaxanthin supplementation among the children with DES. As DES in children is of utmost concern, the current study aims to investigate whether dietary supplementation with astaxanthin could (1) ameliorate the DES symptoms; (2) improve the blue light exposure-associated health complaints; (3) improve the cognitive function and quality of life among the school age children.

ELIGIBILITY:
Inclusion Criteria:

* Children with DES (CVS-Q score 6-18)

Exclusion Criteria:

* Children with CVS-Q score ≥ 19
* Children who wear contact lenses
* Children with any diagnosed ocular motility disorder or accommodative/binocular vision issues
* Participants who are colour-blind
* Participant on any retinols and carotenoid supplements
* Participants who have immunosuppressive disorders or are taking immunosuppressive medication
* Atopy, allergic disorders
* Anaemia
* Ophthalmic laser treatment (less than 3 months)
* Systemic disease associated with dry eye
* Blepharitis
* Having liver (chronic liver failure, cirrhosis, all types of hepatitis), kidney (chronic kidney disease, haemodialysis) or haematological (anaemia, thalassemia, haemophilia) disorders
* Psychiatric disease/mental retardation (bipolar disorder, depression, schizophrenia)
* Cancer (all types), and endocrine disorders (Cushing's disease, gigantism and hyperthyroidism)
* Use of steroids, chemotherapy or radiotherapy
* Currently under another supplementary program

Ages: 10 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Change in Computer Vision Syndrome-Questionnaire score | Baseline, 12 weeks and 24 weeks
  Higher scores mean a worse outcome. The minimum score is 0, while the maximum score is 32

CONTACTS AND LOCATIONS:
Overall Officials: Lai Kuan Dr., PhD, Principal Investigator — Universiti Sains Malaysia
Locations (1):
- Universiti Sains Malaysia Bertam Medical Center, Kepala Batas, Pulau Pinang, Malaysia

IPD SHARING:
Plan to Share IPD: No
Participants are children and they are categorized as vulnerable group.

REFERENCES:
- [Background] Chawla A, Lim TC, Shikhare SN, Munk PL, Peh WCG. Computer Vision Syndrome: Darkness Under the Shadow of Light. Can Assoc Radiol J. 2019 Feb;70(1):5-9. doi: 10.1016/j.carj.2018.10.005. PMID 30691563